CLINICAL TRIAL: NCT01019239
Title: Laparoscopic Lavage for Acute Non-Faeculant Diverticulitis
Brief Title: LapLAND Laparoscopic Lavage for Acute Non-Faeculant Diverticulitis
Acronym: LapLAND
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: St Vincent's University Hospital, Ireland (Other)
Responsible Party: Professor Des C Winter, St. Vincent's University Hospital, Elm Park, Dublin 4.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LapLAND
Record Dates: First submitted 2009-11-23; First posted 2009-11-25 (Estimated); Last update posted 2009-12-01 (Estimated); Status verified 2009-11

CONDITIONS: Diverticulitis
Keywords: Non-faeculant; Perforated; Diverticulitis
MeSH Terms: conditions — Diverticulitis | interventions — Anastomosis, Surgical

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laparoscopic Washout (Experimental): Two 5mm ports will be placed in the suprapubic and right lower quadrants to facilitate triangulation of instruments during manipulation and lavage. The peritoneal cavity will be thoroughly examined and stage classified according to Hinchey. Peritoneal lavage will be performed in all four quadrants using at least 4 litres of warmed saline until the drainage is clear. Two non-suction Penrose drains will be placed. Intravenous antibiotics will be continued for a minimum of 72hours and oral antibiotics will be continued for one week. Oral fluids will be commenced on the first postoperative day and diet will be introduced subsequently, depending on clinical status. Early mobilisation will be encouraged.
  Interventions: Procedure: Laparoscopic Washout
- Conventional Treatment (Active Comparator): Operative procedure will be similar to that previously described.Patients randomised to the second arm will undergo standard management (according to local preference) which will consist of Hartmanns Procedure or Primary resection of the diseased segment and anastomosis. Post operative care will be standardised between arms as described in the protocol
  Interventions: Procedure: Hartmann's Procedure/ Primary Resection and Anastomosis

INTERVENTIONS:
Procedure: Laparoscopic Washout — Pneumoperitoneum will be established via a blunt entry 12mm umbilical port. Two 5mm ports will be placed in the suprapubic and right lower quadrants. The peritoneal cavity will be thoroughly examined and stage classified according to Hinchey. Peritoneal lavage will be performed in all four quadrants using at least 4 litres of warmed saline until the drainage is clear. Two non-suction Penrose drains will be placed.
  Arms: Laparoscopic Washout
Procedure: Hartmann's Procedure/ Primary Resection and Anastomosis — 24 Pneumoperitoneum will be established via a blunt entry 12mm umbilical port. Two 5mm ports will be placed in the suprapubic and right lower quadrants to facilitate triangulation of instruments during manipulation and lavage. The peritoneal cavity will be thoroughly examined and stage classified according to Hinchey. . In the absence of faeculant peritonitis, patients will be randomised to undergo Hartmann's procedure or primary resection and anastomosis (depending on standard practice in the individual unit).
  Arms: Conventional Treatment

SUMMARY:
The aim of the study is to compare patient outcome following standard of care (Hartmann's or resection with anastomosis and defunctioning stoma) and a 'new therapy' (laparoscopic lavage alone) for the treatment of acute perforated non-faeculant diverticulitis in Irish hospitals.

Perforated diverticulitis requires emergency surgery. This carries significant risks and mortality as high as 15% during the index admission has been reported. Our group has established the safety of laparoscopic lavage alone on the largest cohort to date in a prospective multi-institutional study of 100 patients, providing convincing evidence that laparoscopic lavage alone is a reasonable alternative to resection for non-faeculant perforated diverticulitis. Our aim now is to translate this well-established study design into a protocol for a multi-institutional randomised control trial as direct comparison is the only way to provide convincing evidence of one modality over another.

All patients will be followed up for twelve months and primary (operative and in-hospital mortality) and secondary (in-hospital and post-discharge morbidity; rates of stoma formation; rates of re-presentation with diverticulitis with or without perforation.) end-points will be recorded.

Sample size calculations reveal that a patient cohort of 100 in each arm will be sufficient to detect a difference in morbidity and mortality between groups The ratio between Hinchey 3 and Hinchey 4 is estimated to be approximately 2:1. In order to guarantee sufficient sample size, therefore, 300 patients must fulfil the study criteria allowing for exclusion of 100 at time of operation

DETAILED DESCRIPTION:
Background and Current Knowledge:

Until recently, the natural history of diverticular disease was poorly understood and evidence suggesting a link between recurrent presentations with diverticulitis and perforation is almost forty years old rendering its relevance to modern day practice questionable at best . More recently, these questions have been clarified and it seems that risk of perforation following a single (treated) episode of diverticulitis is in the order of 2% per year with a risk of requiring an emergency Hartmann's procedure in this cohort being 1 in 2000 patient years of follow-up . As with all surgical interventions, there is a certain risk profile associated with elective resection and morbidity is estimated at 25-50% (including stoma formation in 10-14%) and mortality at 1-2% . The current vogue (despite some dissention ) is towards a more conservative approach to management of non-perforated acute diverticulitis and away from elective sigmoid colectomy in the absence of perforation .

Management of perforated diverticulitis continues to evolve. The last 50 years has seen standard of care shift from a three stage procedure (1.Drainage and defunctioning colostomy, 2.Excision of diseased segment, 3.Colostomy reversal and restoration of continuity) , to Hartmann's procedure , to resection and primary anastomosis , to treatment with antimicrobial therapy alone in a carefully selected (Hinchey Grade 2) population . Since the learning curve for laparoscopic surgery has begun to plateau, resections for perforated diverticular disease have been shown to be as safe and effective as conventional open techniques .

Irish surgeons have pioneered the institution of laparoscopic lavage for acute non-faeculant diverticulitis. The operative method described involves laparoscopy, copious washout, drain placement and treatment with antimicrobial therapy (intravenous for 72hours followed by oral for one week). Benefits include low mortality, stoma avoidance, minimal wound infection, shorter operative time and no difference in recurrence when compared to primary resection and anastomosis. Having demonstrated a clear clinical advantage of laparoscopic lavage over standard of care (Hartmann's procedure or primary resection and anastomosis) for acute non faeculant perforated diverticulitis, we feel the time is ripe to formalise these findings through performance of a multicentre national randomised controlled trial- LapLAND (LAParoscopic Lavage for Acute Non-faeculant Diverticulitis).

Relevance:

Perforated diverticulitis requires emergency surgery . This carries significant risks and mortality as high as 15% during the index admission has been reported . It appears that morbidity and mortality related to resections in complicated and uncomplicated disease are reduced in laparoscopic intervention when compared to open . The real question, however, is whether or not there is necessity to perform any resection or whether lavage is sufficient. Our group has established the safety of this procedure on the largest cohort to date24 in a prospective multi-institutional study of 100 patients. We provided convincing evidence that laparoscopic lavage is a reasonable alternative to resection for non-faeculant perforated diverticulitis. We demonstrated a low mortality rate despite patient co-morbidity and disease severity. Benefits of lavage alone included stoma avoidance and decreased wound infection. At up to 36 months follow up it appeared that subsequent resection appeared unnecessary. These findings were confirmed by a similar French trial published this year which demonstrated no excess morbidity or mortality, a reduction in hospital stay and a lower rate of stoma formation. Having established the safety of the new intervention (laparoscopic lavage), our aim now is to translate this well established study design into a protocol for a multi-institutional randomised control trial as we believe that direct comparison is the only way to provide convincing evidence of one modality over another.

Knowledge transfer/implementation/consolidation:

Evidence to date regarding the management of perforated diverticulitis is based on a combination of eminence based opinion and outdated retrospective analysis. A true prospective analysis comparing standard of care (Hartmann's or resection with anastomosis and defunctioning stoma) and a 'new therapy' (laparoscopic lavage alone) is yet to be published. Aims and Objective:

To compare patient outcome following standard of care (Hartmann's or resection with anastomosis and defunctioning stoma) and a 'new therapy' (laparoscopic lavage alone) for the treatment of acute perforated non-faeculant diverticulitis in Irish hospitals. Specific research questions include:

1. Which treatment modality confers least mortality and morbidity in patients with non-faeculant perforated diverticulitis?
2. Does treatment influence length of hospital stay and return to activities of daily living?
3. Do patients undergoing laparoscopic lavage alone require emergency sigmoidectomy at a later date (within a one year period)?
4. Does laparoscopic lavage alone confer any advantage in terms of stoma-free survival?

Strategy:

An Irish multi-centre trial will be performed with the aim of comparing two treatment modalities for patients presenting acutely with perforated non-faeculant diverticulitis. Pre-operative details, intraoperative findings and post-operative course will be prospectively accrued by the operating surgeon. All patients will be followed up for twelve months and primary (operative and in-hospital mortality) and secondary (in-hospital and post-discharge morbidity; rates of stoma formation; rates of re-presentation with diverticulitis with or without perforation.) end-points will be recorded.

Study Outline:

All patients demonstrating clinical signs of generalised peritonitis and radiological evidence of intra-peritoneal free air (on erect chest radiograph or abdominal CT scan will be eligible for the study. Individual patient consent will be sought. They will be given intravenous fluids (standardised regime) and intravenous antibiotics (3rd generation cephalosporin and metronidazole). All patients will be given prophylaxis against deep vein thrombosis (compression stockings and low molecular weight heparin). When patients have received adequate fluid resuscitation they will proceed to theatre on an emergency basis.

Pneumoperitoneum will be established via a blunt entry umbilical port. Two 5mm ports will be placed in the suprapubic and right lower quadrants to facilitate triangulation of instruments during manipulation and lavage. The peritoneal cavity will be thoroughly examined and stage classified according to Hinchey. All patients with faeculant peritonitis will undergo Hartmann's procedure or primary resection and anastomosis according to local preference and excluded from the study on that basis. In the absence of faeculant peritonitis, patients will be randomised to undergo Hartmann's procedure or primary resection and anastomosis (depending on standard practice in the individual unit) or laparoscopic lavage alone. Peritoneal lavage will be performed in all four quadrants using at least 4 litres of warmed saline until the drainage is clear. Intravenous antibiotics will be continued for a minimum of 72hours and oral antibiotics will be continued for one week. Oral fluids will be commenced on the first postoperative day and diet will be introduced subsequently, depending on clinical status. Early mobilisation will be encouraged.

Study Management:

This multicentre surgical clinical trial will be coordinated by the R&D unit of the Colles Institute at RCSI. The Colles Institute comprises of the National Surgical Training Centre, the Centre of R&D and Centre for Innovation in Surgical Technology. The Project Manager for this trial will be Mr Kieran Ryan, who has over 10 years experience in running clinical trials along with many years experience in the Irish Health System, including his role as a former GCP inspector with the Irish Medicines Board. Kieran and his team will ensure that the trial is carried out in accordance with the relevant regulations, GCP standards and the requirements of the protocol. This will ensure the smooth running of the trial and the integrity of the research data and management of the patients.

There will also be a DSMB (Data & Safety Monitoring Board) of external surgeons established to oversee the progress of the study and ensure that the safety of patients are to the forefront of this trial.

Data Collection:

Data collection will be performed by the operating surgeon or a designated member of the surgical team (present at time of operation) and recorded on an electronic pro-forma or electronic Case Report Form. It will include patient demographics (age, sex), previous diverticular history American Society of Anaesthesiologists (ASA) grade and specific co-morbidities, intervention performed, operation performed, incidence of stoma formation, re-intervention during index admission (radiological or operative) in-hospital morbidity (myocardial infarction, deep vein thrombosis, pulmonary embolism, wound infection, abscess requiring drainage, urosepsis, renal failure or respiratory insufficiency), mortality, time to return to diet, time to discharge. Further details will be recorded at post-operative visits- stoma-free survival at one year, number of days alive following discharge, reinterventions within 12 months, patient satisfaction.

Standardisation of treatment within trial:

Patients may withdraw from the trial at any time if they so wish. Re-laparotomy may be performed at the discretion of the operating surgeon but fixed indications include clinical deterioration or failure to improve within 48-72 hours post-operatively. Potential foci of concurrent sepsis should be out-ruled (respiratory, urinary) by clinical, biochemical or radiological investigations.

Hospital Inclusion and Patient Accrual:

All eligible patients (see exclusion criteria) presenting to participating hospitals with perforated diverticulitis will be recruited for the trial. They will be furnished with a patient information leaflet and will have the implications of inclusion in the trial explained to them by the operating surgeon. It will be explained that non-willingness to participate in the trial will not have any negative impact on their treatment. If the patient is willing to participate in the trial, verbal and written consent will be obtained prior to transfer to the operating theatre.

Sample size Calculation:

Having performed an extensive literature review of studies comparing treatment entities for perforated non-faeculant diverticulitis, sample size calculations reveal that a patient cohort of 100 in each arm will be sufficient to detect a difference in morbidity and mortality between groups (25% versus 10%; two sided significance 5% and a power of 80%). A significance level of 0.05 on the two sided Likelihood ratio test was used and the significance level achieved by this design is 0.04997.

In order to guarantee sufficient sample size, therefore, 300 patients must fulfil the study criteria (allowing for exclusion of 100 at time of operation). Recruitment of patients is not expected to be difficult because evidence to date is convincing of at least equivalent outcome and we believe that most patients would hope to be assigned to the lavage group in the hope of avoiding a stoma. From a surgeon's perspective, laparoscopic lavage is technically less challenging and time consuming than traditional treatment modalities.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-85 years..
2. Clinical evidence of generalised peritonitis.
3. Free air on erect chest x-ray or CT abdomen suggestive of perforated diverticulitis.
4. Informed consent.

Exclusion Criteria:

1. Inability to give informed consent (eg dementia).
2. Prior sigmoidectomy.
3. Ongoing steroid treatment >20mg/day.
4. Prior pelvic irradiation.
5. Requirement for inotropic support pre-operatively.
6. Faecal peritonitis or overt sigmoid perforation (demonstrated on laparoscopy).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2010-01; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Operative and in-hospital mortality | 1 year

SECONDARY OUTCOMES:
In-hospital and post-discharge morbidity | 1 year
Rates of stoma formation | 1 year
Rates of re-presentation with diverticulitis with or without perforation | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Aisling M Hogan, MD, Study Director — St Vincent's University Hospital, Ireland; Kieran Ryan, BSc, Study Director — Royal College of Surgeons in Ireland; Des C Winter, MD, Principal Investigator — St Vincent's University Hospital and Royal College of Surgeons in Ireland
Locations (1):
- Royal College of Surgeons in Ireland, Dublin, Dublin, Ireland

REFERENCES:
- [Background] Karoui M, Champault A, Pautrat K, Valleur P, Cherqui D, Champault G. Laparoscopic peritoneal lavage or primary anastomosis with defunctioning stoma for Hinchey 3 complicated diverticulitis: results of a comparative study. Dis Colon Rectum. 2009 Apr;52(4):609-15. doi: 10.1007/DCR.0b013e3181a0a674. PMID 19404062
- [Background] Myers E, Hurley M, O'Sullivan GC, Kavanagh D, Wilson I, Winter DC. Laparoscopic peritoneal lavage for generalized peritonitis due to perforated diverticulitis. Br J Surg. 2008 Jan;95(1):97-101. doi: 10.1002/bjs.6024. PMID 18076019
- [Background] O'Sullivan GC, Murphy D, O'Brien MG, Ireland A. Laparoscopic management of generalized peritonitis due to perforated colonic diverticula. Am J Surg. 1996 Apr;171(4):432-4. doi: 10.1016/S0002-9610(97)89625-0. PMID 8604837
- [Background] Collins D, Winter DC. Elective resection for diverticular disease: an evidence-based review. World J Surg. 2008 Nov;32(11):2429-33. doi: 10.1007/s00268-008-9705-7. PMID 18712563
- [Derived] Rogers AC, Collins D, O'Sullivan GC, Winter DC. Laparoscopic lavage for perforated diverticulitis: a population analysis. Dis Colon Rectum. 2012 Sep;55(9):932-8. doi: 10.1097/DCR.0b013e31826178d0. PMID 22874599